CLINICAL TRIAL: NCT07276672
Title: Efficacy of a Toothpaste Containing Hydrogen Peroxide as Compared to a Regular Fluoride Toothpaste Without Hydrogen Peroxide in the Immediate Removal of Tooth Stains After a Single Brushing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-07-STN-OW2-DR-BGS
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Whitening
Keywords: Hydrogen Peroxide
MeSH Terms: interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 toothpaste (Experimental): 2%HPToothpaste
  Interventions: Drug: Optic White Adv Sparkling White (2%HP) Toothpaste
- Test 2 toothpaste (Active Comparator): .76% Na MFP toothpaste
  Interventions: Drug: Colgate Great Regular Flavor Toothpaste

INTERVENTIONS:
Drug: Optic White Adv Sparkling White (2%HP) Toothpaste — 0.243% NaF toothpaste
  Arms: Test 1 toothpaste
Drug: Colgate Great Regular Flavor Toothpaste — 0.76% Na MFP
  Arms: Test 2 toothpaste

SUMMARY:
The aim of this study is to evaluate and compare the immediate efficacy of a hydrogen peroxide-containing toothpaste versus a regular fluoride toothpaste without hydrogen peroxide in removing extrinsic tooth stains following a single supervised brushing in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Male and female subjects, aged 18-70, inclusive;
* Good general health and good oral health based on the opinion of the study investigator; - Presence of permanent natural anterior teeth (no veneers/crowns/restorations that may interfere with this study scoring procedures);
* A minimum composite mean of ≥ 1.5 determined by the Mod. Lobene Tooth Stain Index;
* Available for the duration of the study;
* Clinical evidence of a tendency to form extrinsic stains on anterior teeth

Exclusion Criteria:

* Presence of orthodontic appliances/retainers involving scorable teeth;
* Presence of partial removable/fixed dentures and/or restorations involving scorable teeth; 3. Tumor(s) of the soft or hard tissues of the oral cavity;
* Obvious signs of periodontal disease rampant caries, or any condition that the dental examiner considers exclusionary from the study;
* Five or more carious lesions requiring immediate care;
* Use of antibiotics, stain-inducing medications, and/or on any prescription that might interfere with the study outcome;
* Concurrent participation in another clinical study;
* Self-reported pregnancy and/or lactating women;
* Have used professional whitening product within one (1) year or had a dental prophylaxis (professional dental cleaning) within thirty (30) days - prior to the start of the study
* History of allergies or sensitivity to tooth whitening products, hydrogen peroxide, personal care consumer products, or their ingredients;
* History of alcohol and/or drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Mod. Lobene Stain Index | one day
  each tooth will be scored separately using a 4 point area and intensity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Spa Dental, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No